CLINICAL TRIAL: NCT01865279
Title: A Randomised, Double-blind, Placebo-controlled Single Dose, Dose Escalation Trial With Insulin 454 in Healthy Male Subjects, Followed by a Two-period Cross-over Trial With Insulin 454 and Insulatard® in Male Subjects With Type 1 and Type 2 Diabetes Mellitus
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Explorative Formulation of Insulin Degludec
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN5401-1718; 2005-003974-65 (EudraCT Number)
Record Dates: First submitted 2013-05-27; First posted 2013-05-30 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin, Isophane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trial part 1 (Experimental)
  Interventions: Drug: insulin degludec; Drug: placebo
- Trial part 2 (Active Comparator)
  Interventions: Drug: insulin degludec; Drug: isophane human insulin

INTERVENTIONS:
Drug: insulin degludec — Ascending single doses - 5 dose levels. Escalation to next dose level will be performed following evaluation of safety data.
  Arms: Trial part 1
Drug: placebo — Ascending single doses - 5 dose levels
  Arms: Trial part 1
Drug: insulin degludec — A single dose corresponding to that of isophane human insulin
  Arms: Trial part 2
Drug: isophane human insulin — A single dose of 0.4 IU/kg is administered to subjects with type 1 diabetes while a single dose of 0.6 IU/kg is administered to subjects with type 2 diabetes
  Arms: Trial part 2

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the safety, tolerability, pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of insulin degludec (insulin 454), an explorative formulation, not similar to the proposed commerical formulation.

ELIGIBILITY:
Inclusion Criteria:

* HEALTHY SUBJECTS:
* Subjects will be healthy male subjects, who are considered to be generally healthy based on an assessment of medical history, physical examination and clinical laboratory data, as judged by the Investigator
* Body mass index (BMI) between 18.0-27.0 kg/m^2 (both inclusive)
* SUBJECTS WITH TYPE 1 AND TYPE 2 DIABETES:
* Subjects will be male volunteers, who are considered to be generally healthy, except for the underlying diabetes mellitus, based on an assessment of medical history, physical examination and clinical laboratory data, as judged by the Investigator
* Diagnosed with type 1 diabetes mellitus and treated with insulin for at least 12 months or diagnosed with type 2 diabetes mellitus for at least 12 months
* Body Mass Index (BMI) between 18.0-27.0 kg/m^2 (both inclusive) for subjects with type 1 diabetes or 25.0-35.0 kg/m^2 (both inclusive) for subjects with type 2 diabetes
* Glycogylated haemoglobin (HbA1c) maximum 8.5 % based on central laboratory results
* Subjects with type 2 diabetes must have been treated with insulin for the past 3 months prior to screening

Exclusion Criteria:

* Participation in any other trials involving investigational products within 3 months preceding the start of dosing
* History of significant multiple drug allergies or with a known allergy to the trial product or any medicine chemically related to the trial product, as judged by the investigator
* Hepatitis or carrier of the Hepatitis B surface antigen (HBsAg) or Hepatitis C antibodies or a positive result to the test for human immunodeficiency (HIV) antibodies
* Any clinically significant abnormal haematology or biochemistry screening tests, as judged by the investigator
* Subjects who have donated any blood or plasma in the past month or in excess of 1000 ml within the 12 weeks preceding screening

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2005-12; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (trial part 1 only) | From day prior to dosing and until 10-14 days after dosing
Area under the glucose infusion rate curve (trial part 2 only) | 0-24 hours after dosing

SECONDARY OUTCOMES:
Area under the serum insulin concentration curve | 0-72 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com